CLINICAL TRIAL: NCT07049887
Title: A Multicenter Non-interventional Study for the Measurement of Scratch and Sleep Patterns Using the ADAM Sensor in Patients With Primary Biliary Cholangitis
Brief Title: A Study Describing Scratch and Sleep Patterns in Patients With Primary Biliary Cholangitis (Luminaria)
Status: Active, not recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60190-466
Record Dates: First submitted 2025-06-09; First posted 2025-07-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will collect information from patients with Primary Biliary Cholangitis (PBC).

PBC is a progressive rare liver disease in which tubes in the liver called bile ducts are damaged. The liver damage in PBC may lead to scarring (cirrhosis). People living with PBC often face challenges like intense itching, trouble sleeping, and feeling constantly tired. These symptoms can make it hard for them to enjoy daily life and feel well overall.

While itching and sleep patterns can be difficult to measure accurately based on recall and may lack precision, the main aim of this study is to use a digital health tool to assess the severity of itchiness and sleep patterns in people with PBC. The tool will take the objective measurement for people so they do not have to recall their scratch and sleep patterns. The total study duration for each patient will be about 91 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at time of study enrollment.
* Confirmed diagnosis of PBC based on medical history and relevant clinical criteria, as determined by the study Investigator.
* Willingness and ability to wear the ADAM sensor during the specified time periods (7 nights across four 7-day periods).
* Able to read and write to ensure accurate completion of electronic PRO surveys.
* Able to access an internet-connected device for the completion of electronic PRO surveys.
* Able to provide signed, informed consent prior to collection of data.

Exclusion Criteria:

* Has already been enrolled in another clinical study.
* Has any dermatological conditions or severe comorbidities associated with pruritus as assessed by the investigators that may confound the measurement of scratch or sleep data.
* Has any extrapyramidal syndrome including Parkinsonism, essential tremor, astasia/abasia, cerebellar syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with PBC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Nocturnal Scratch Events | At weeks 0, 4, 8 and 12
  Defined as the total number of scratch events detected during sleep periods, monitored using the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Frequency of Low- and High-Intensity Nocturnal Scratch Events | At weeks 0, 4, 8 and 12
  Defined as the frequency of scratch events categorized into low- and high-intensity levels during sleep periods, as detected by the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Average Scratch Intensity Per Night | At weeks 0, 4, 8 and 12
  Defined as the average intensity of scratch events per night, calculated from data recorded by the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Hourly Frequency of Nocturnal Scratch Events During Sleep | At weeks 0, 4, 8 and 12
  Defined as the frequency of nocturnal scratch events occurring per hour during sleep periods, recorded using the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Average Duration of Scratch Events Per Night | At weeks 0, 4, 8 and 12
  Defined as the average duration of scratch events occurring during sleep periods, calculated using data collected via the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Total Duration of Scratch Behavior Per Patient During Sleep Periods | At weeks 0, 4, 8 and 12
  Defined as the total duration of scratch events recorded for each patient during sleep periods using the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Total Sleep Duration (Hours) | At weeks 0, 4, 8 and 12
  Defined as the total duration of sleep per patient, recorded by the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Duration of Wakefulness After Sleep Onset (WASO, Minutes) | At weeks 0, 4, 8 and 12
  Defined as the total duration of wakefulness after the initial onset of sleep, measured using the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Duration of Wakefulness During Scratch Periods | At weeks 0, 4, 8 and 12
  Defined as the total duration of wakefulness during scratch periods, monitored via the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.
Average Sleep Duration Between Scratch Periods | At weeks 0, 4, 8 and 12
  Defined as the average duration of sleep occurring between scratch periods, as measured by the Nighttime sensor wear. This outcome will be assessed at the end of the wear period.

SECONDARY OUTCOMES:
Demographic Data: Age at Enrollment | At enrollment visit (Week 0, Day 1)
  Defined as the age of patients recorded at the time of enrollment.
Demographic Data: Sex at Enrollment | At enrollment visit (Week 0, Day 1)
  Defined as the sex of patients recorded at the time of enrollment.
Age at Diagnosis (As Available) | At enrollment visit (Week 0, Day 1)
  Defined as the patient's age at the time of diagnosis, as reported in their medical history.
Age at First Symptoms (As Available) | At enrollment visit (Week 0, Day 1)
  Defined as the patient's age when first symptoms were reported, based on medical records or patient recollection.
Time Duration Since PBC Diagnosis | At enrollment visit (Week 0, Day 1)
  Defined as the duration between the patient's initial diagnosis of PBC and the time of enrollment, as recorded in their medical history.
Current PBC-Related Treatments | At enrollment visit (Week 0, Day 1)
  Defined as the treatments patients are currently receiving for PBC, including medication and other therapies, as reported at enrollment.
Time Duration on Current PBC-Related Treatment | At enrollment visit (Week 0, Day 1)
  Defined as the duration for which patients have been receiving their current PBC-related treatment, as recorded during enrollment.
Concomitant Medications for Itch/Scratch and/or Sleep Disturbances | At enrollment visit (Week 0, Day 1)
  Defined as the additional medications patients are currently using to manage itch/scratch and/or sleep disturbances, as reported at enrollment.
Baseline Liver Function Tests: Alanine aminotransferase (ALT) Levels | At enrollment visit (Week 0, Day 1)
Baseline Liver Function Tests: Aspartate aminotransferase (AST) Levels | At enrollment visit (Week 0, Day 1)
Baseline Liver Function Tests: Alkaline phosphatase (ALP) Levels | At enrollment visit (Week 0, Day 1)
Baseline Liver Function Tests: Bilirubin Levels | At enrollment visit (Week 0, Day 1)
Baseline Liver Function Tests: Albumin Levels | At enrollment visit (Week 0, Day 1)
Baseline Enhanced Liver Fibrosis (ELF) Test: Hyaluronic Acid (HA) Levels | At enrollment visit (Week 0, Day 1)
Baseline ELF Test: Procollagen Type III Amino-Terminal Propeptide (PIIINP) Levels | At enrollment visit (Week 0, Day 1)
Baseline ELF Test: Tissue Inhibitor of Metalloproteinase-1 (TIMP-1) Levels | At enrollment visit (Week 0, Day 1)
Baseline Liver Stiffness Measurement by Fibroscan | At enrollment visit (Week 0, Day 1)
PBC Worst Itch Numeric Rating Scale (PBC WI NRS) Score | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the PBC WI NRS, assessing the severity of worst itch experienced during the study duration.
PBC-40 Itch Severity Score | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the itch severity domain of the PBC-40 questionnaire, measuring the impact of itch on their quality of life.
Duration, degree, direction, disability, and distribution (5-D) Itch Scale | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the 5-D Itch Scale, capturing dimensions of duration, degree, direction, disability, and distribution of itch.
PBC-40 Fatigue Severity Score | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the fatigue severity domain of the PBC-40 questionnaire, quantifying the impact of fatigue on their daily life.
Sleep Disturbance Numeric Rating Scale (SD NRS) Score | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the SD NRS, evaluating the severity of sleep disturbances experienced during the study duration.
Patient-Reported Outcomes Measurement Information System® (PROMIS®) Fatigue Short Form (SF)-7a Score | At weeks 0, 4, 8 and 12
  Defined as the patient's score on the PROMIS® Fatigue SF-7a, assessing fatigue levels and their effects on physical, mental, and social activities.
Percentage of Patient Responses to Sibel Health System Usability Survey (SUS) | At week 12 (End of Study Survey)
  Defined as the patients' feedback on the usability of the Sibel Health System, captured through the SUS administered during enrollment. This outcome will assess user experience and satisfaction with the system.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- United States (3):
  - Arizona Liver Center, Chandler, Arizona
  - University of Miami School of Medicine, Center for Liver Diseases, Miami, Florida
  - UT Southwestern Medical Center, Department of Internal Medicine, Digestive and Liver Diseases, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency